CLINICAL TRIAL: NCT00057018
Title: The Extremity Constraint Induced Therapy Evaluation (EXCITE) Trial
Brief Title: Improving Arm Mobility and Use After Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD037606 (NIH)
Record Dates: First submitted 2003-03-26; First posted 2003-03-28 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2011-05

CONDITIONS: Cerebrovascular Accident
Keywords: stroke; cerebrovascular accident; upper extremity; physical therapy; constraint-induced therapy
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy

INTERVENTIONS:
Procedure: Constraint-induced movement therapy

SUMMARY:
An individual suffering a stroke or other brain injury may lose function on one side of the body (partial paralysis). As the individual shifts activities to favor the unaffected side, the problem worsens. Constraint induced (CI) therapy forces the individual to use the neglected arm by restraining the good arm in a sling. This study examines the effectiveness of CI therapy for improving arm motion after stroke.

DETAILED DESCRIPTION:
Profoundly impaired motor dysfunction is a major consequence of stroke. As a result, a large number of the more than 700,000 people in America sustaining a stroke each year have limitations in motor ability and compromised quality of life. Therapeutic interventions designed to enhance motor function and promote independent use of an impaired upper extremity are quite limited.

CI movement therapy, or "forced use," involves motor restriction of the less effected upper extremity for 2 weeks. Over this time, repetitive use of the more effected upper extremity is promoted for many hours a day. This treatment produces long lasting improvements in extremity use among patients who are more than 1 year post-stroke and who have an ability to initiate some extension in wrist and digit joints.

This study will determine if CI therapy for a hemiparetic upper extremity in patients with sub-acute (3 to 9 months post-cerebral infarct) stroke will lead to functional improvements and enhanced quality of life measures more than usual care.

Patients are randomized into a treatment or usual care group and stratified by movement capability into higher and lower functioning categories. Higher functioning patients are defined as those who have at least 20 degrees of active wrist extension and 10 degrees of active finger extension at each digit joint. Lower functioning patients are defined as those with at least 10 degrees of wrist extension and 10 degrees of extension at each thumb joint and all joints of two other digits. Patients randomized into the control group receive treatment one year later to permit replication efforts for findings using this therapy in patients with chronic stroke.

The intervention consists of making patients use their impaired arms by constraining movement in the less impaired limb for most waking hours over a 2 week period. The constraint is a taped splint in which the hand rests to prevent limb use but enable protective responses. A micro-switch within the splint will permit monitoring of contact time (wearing). Each weekday for 2 weeks, patients come to the clinic/laboratory for specific task training. Evaluations in laboratory and actual use tests are made prior to treatment, 2 weeks later, and at 4 month intervals thereafter. Changes in psychosocial functioning will also be measured. Primary outcomes include the Wolf Motor Function Test and the Motor Activity Log. Secondary outcomes include Stroke Impact Scale, Actual Amount of Use Test, and accelerometry.

ELIGIBILITY:
Inclusion Criteria

* 3 to 9 months post cerebral infarct or 1 year post injury
* 2.5 or lower on the Motor Activity Log scale
* >= 10 degrees of active wrist extension
* >= 10 degrees of extension of all joints of thumb and two other digits
* Ability to perform wrist/finger extension movements three times within one minute

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229
Dates: Start 2000-04; Primary Completion 2005-03 (Actual); Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Wolf, PhD/PT/FAPTA, Principal Investigator — Emory University
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Ostendorf CG, Wolf SL. Effect of forced use of the upper extremity of a hemiplegic patient on changes in function. A single-case design. Phys Ther. 1981 Jul;61(7):1022-8. doi: 10.1093/ptj/61.7.1022. PMID 7243897
- [Background] Wolf SL, Lecraw DE, Barton LA, Jann BB. Forced use of hemiplegic upper extremities to reverse the effect of learned nonuse among chronic stroke and head-injured patients. Exp Neurol. 1989 May;104(2):125-32. doi: 10.1016/s0014-4886(89)80005-6. PMID 2707361
- [Background] Taub E, Crago JE, Burgio LD, Groomes TE, Cook EW 3rd, DeLuca SC, Miller NE. An operant approach to rehabilitation medicine: overcoming learned nonuse by shaping. J Exp Anal Behav. 1994 Mar;61(2):281-93. doi: 10.1901/jeab.1994.61-281. PMID 8169577
- [Background] Taub E: Somatosensory deafferentation research with monkeys: Implications for rehabilitation medicine. In Ince LP (ed.) Behavioral Psychology in Rehabilitation Medicine: Clinical Applications. New York: Williams Wilkins, 1980, 370-401
- [Background] Taub E, Miller NE, Novack TA, Cook EW 3rd, Fleming WC, Nepomuceno CS, Connell JS, Crago JE. Technique to improve chronic motor deficit after stroke. Arch Phys Med Rehabil. 1993 Apr;74(4):347-54. PMID 8466415
- [Background] Taub E, Pidikiti RD, DeLuca SC, Crago JE: Effects of motor restriction of an unimpaired upper extremity and training on improving functional tasks and altering brain/behaviors. In J. Toole (ed.), Imaging and Neurologic Rehabilitation. New York::Demos, 1996, 133-154.
- [Background] Taub E, Wolf SL. Constraint Induced Movement Techniques To Facilitate Upper Extremity Use in Stroke Patients. Top Stroke Rehabil. 1997 Jan;3(4):38-61. doi: 10.1080/10749357.1997.11754128. PMID 27620374
- [Background] Taub E, Morris DM. Constraint-induced movement therapy to enhance recovery after stroke. Curr Atheroscler Rep. 2001 Jul;3(4):279-86. doi: 10.1007/s11883-001-0020-0. PMID 11389792
- [Background] Duncan PW. Synthesis of Intervention Trials To Improve Motor Recovery following Stroke. Top Stroke Rehabil. 1997 Jan;3(4):1-20. doi: 10.1080/10749357.1997.11754126. PMID 27620372
- [Background] Wolf SL, Blanton S, Baer H, Breshears J, Butler AJ. Repetitive task practice: a critical review of constraint-induced movement therapy in stroke. Neurologist. 2002 Nov;8(6):325-38. doi: 10.1097/01.nrl.0000031014.85777.76. PMID 12801434
- [Background] Clark PC, Shields CG, Aycock D, Wolf SL. Preliminary reliability and validity of a family caregiver conflict scale for stroke. Prog Cardiovasc Nurs. 2003 Spring;18(2):77-82, 92. PMID 12732800
- [Background] Butler AJ, Wolf SL. Transcranial magnetic stimulation to assess cortical plasticity: a critical perspective for stroke rehabilitation. J Rehabil Med. 2003 May;(41 Suppl):20-6. doi: 10.1080/16501960310010106. PMID 12817653
- [Background] Winstein CJ, Miller JP, Blanton S, Taub E, Uswatte G, Morris D, Nichols D, Wolf S. Methods for a multisite randomized trial to investigate the effect of constraint-induced movement therapy in improving upper extremity function among adults recovering from a cerebrovascular stroke. Neurorehabil Neural Repair. 2003 Sep;17(3):137-52. doi: 10.1177/0888439003255511. PMID 14503435
- [Background] Aycock DM, Blanton S, Clark PC, Wolf SL. What is constraint-induced therapy? Rehabil Nurs. 2004 Jul-Aug;29(4):114-5, 121. doi: 10.1002/j.2048-7940.2004.tb00326.x. No abstract available. PMID 15222091
- [Background] Park SW, Butler AJ, Cavalheiro V, Alberts JL, Wolf SL. Changes in serial optical topography and TMS during task performance after constraint-induced movement therapy in stroke: a case study. Neurorehabil Neural Repair. 2004 Jun;18(2):95-105. doi: 10.1177/0888439004265113. PMID 15228805
- [Background] Wolf SL, Butler AJ, Campana GI, Parris TA, Struys DM, Weinstein SR, Weiss P. Intra-subject reliability of parameters contributing to maps generated by transcranial magnetic stimulation in able-bodied adults. Clin Neurophysiol. 2004 Aug;115(8):1740-7. doi: 10.1016/j.clinph.2004.02.027. PMID 15261852
- [Result] Wolf SL, Winstein CJ, Miller JP, Taub E, Uswatte G, Morris D, Giuliani C, Light KE, Nichols-Larsen D; EXCITE Investigators. Effect of constraint-induced movement therapy on upper extremity function 3 to 9 months after stroke: the EXCITE randomized clinical trial. JAMA. 2006 Nov 1;296(17):2095-104. doi: 10.1001/jama.296.17.2095. PMID 17077374
- [Derived] Schweighofer N, Ye D, Luo H, D'Argenio DZ, Winstein C. Long-term forecasting of a motor outcome following rehabilitation in chronic stroke via a hierarchical bayesian dynamic model. J Neuroeng Rehabil. 2023 Jun 29;20(1):83. doi: 10.1186/s12984-023-01202-y. PMID 37386512
- [Derived] Wolf SL, Thompson PA, Winstein CJ, Miller JP, Blanton SR, Nichols-Larsen DS, Morris DM, Uswatte G, Taub E, Light KE, Sawaki L. The EXCITE stroke trial: comparing early and delayed constraint-induced movement therapy. Stroke. 2010 Oct;41(10):2309-15. doi: 10.1161/STROKEAHA.110.588723. Epub 2010 Sep 2. PMID 20814005
- [Derived] Wolf SL, Winstein CJ, Miller JP, Thompson PA, Taub E, Uswatte G, Morris D, Blanton S, Nichols-Larsen D, Clark PC. Retention of upper limb function in stroke survivors who have received constraint-induced movement therapy: the EXCITE randomised trial. Lancet Neurol. 2008 Jan;7(1):33-40. doi: 10.1016/S1474-4422(07)70294-6. PMID 18077218